CLINICAL TRIAL: NCT00152204
Title: Community Effectiveness of Intermittent Preventive Treatment Delivered Through the Expanded Programme of Immunisation for Malaria and Anaemia Control in Tanzanian Infants
Brief Title: The Community Effectiveness of IPTi in Southern Tanzania
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Research and Development Centre (Other); Ministry of Health, Tanzania (Other Government); Hospital Clinic of Barcelona (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: David Schellenberg, London School of Hygiene & Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMGF28580
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Malaria, Falciparum; Anemia
Keywords: Use-Effectiveness; Cost Effectiveness; Patient Acceptance of Health Care; Drug Resistance; Delivery of Health Care
MeSH Terms: conditions — Malaria, Falciparum; Anemia; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Doses of IPTi with SP delivered alongside doses 2 & 3 of DTP/HB vaccination and alongside measles vaccination
  Interventions: Drug: Sulfadoxine-pyrimethamine used for IPTi; Drug: IPTi
- 2 (No Intervention)

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine used for IPTi — Doses of IPTi with SP delivered alongside doses 2 & 3 of DTP/HB vaccination and alongside measles vaccination
  Other Names: Brand of SP used is Fanisdar
  Arms: 1
Drug: IPTi — Doses of IPTi with SP delivered alongside doses 2 & 3 of DTP/HB vaccination and alongside measles vaccination
  Other Names: SP brand being used is Fansidar
  Arms: 1

SUMMARY:
The safety and efficacy of Intermittent Preventive Treatment for malaria and anaemia control in Infants (IPTi) have already been documented in Southern Tanzania, affording an opportunity to gain operational experience in developing a strategy for the longer-term implementation of IPTi. Working in conjunction with national and district-based health authorities, a strategy will be developed to make IPTi available through routine health services and an effectiveness evaluation conducted. This will be based on the comparison of process and outcome indicators in areas with and without IPTi. Information on safety will be consolidated and the effect of IPTi on the rate of development of drug resistance explored. The acceptability and costs of implementing IPTi will be monitored and combined with assessments of effectiveness (in terms of morbidity and mortality) to assess the cost-effectiveness of IPTi.

DETAILED DESCRIPTION:
A controlled trial of intermittent preventive malaria treatment in infants (IPTi) in southern Tanzania showed that treatment doses of antimalarial given to children at the time of routine vaccinations in the first year of life reduced the incidence of clinical malaria by 59% and halved the amount of severe anaemia. There were also useful reductions in presentations to hospital with fever (13%) and admission to hospital (30%). IPTi was safe, did not interfere with the serological response to EPI vaccines, cost approximately US$ 0.23 per child and the drug used (sulphadoxine-pyrimethamine) is readily available in Tanzania. Hence it is possible to reduce the rate of clinical malaria and severe anaemia by delivering an available and affordable drug through the existing EPI system in southern Tanzania.

Under the umbrella of the IPTi Consortium, a number of similar studies are now planned or underway to assess the safety and efficacy of IPTi in different settings and to confirm the non-interaction between various antimalarials used for IPTi and EPI vaccines. The aim is to generate robust information to inform a policy recommendation on the use of IPTi. The challenge will be to transform a positive policy recommendation into public health action in a short timeframe. Southern Tanzania is now in the unique position of being able to address the issues surrounding the development and implementation of IPTi as part of a district-based strategy to control malaria.

This project will develop, implement and evaluate a strategy for the delivery of IPTi to communities in five rural districts in southern Tanzania. IPTi will be delivered by routine health services in half of the facilities in the project area. Comparison of process and outcome indicators in areas with and without the IPTi strategy will provide an opportunity to consolidate the safety profile of IPTi and to evaluate its impact on (i) the rate of development of antimalarial drug resistance, (ii) perceptions and compliance with the EPI programme and (iii) infant health and survival patterns. The effectiveness evaluation will be linked to costing data to produce realistic estimates of cost effectiveness of the IPTi strategy.

ELIGIBILITY:
Inclusion Criteria:

* child attending routine vaccination services for second or third dose of diptheria/pertussis/tetanus vaccinations (aged approximately two and three months, respectively) or for measles vaccination (aged approximately 9 months)

Exclusion Criteria:

* sensitivity to sulfadoxine-pyrimethamine or other sulfur-containing drugs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13000 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate in children aged 2-11 months (estimated by birth history questioning) | Up to 12 months of age
Incidence of severe adverse drug reactions following IPTi (as detected by spontaneous, passive reporting system) | All age groups, particular attention in under 2 year olds

SECONDARY OUTCOMES:
Prevalence of P falciparum parasitemia in children aged 2-11 months. | First year of life
Prevalence of anaemia (Hb<11 g/dL) in children aged 2-11 months. | First year of life
Period prevalence of fever without cough or diarrhoea (in preceding 2 weeks) in children aged 2-11 months. | First year of life

CONTACTS AND LOCATIONS:
Overall Officials: David M Schellenberg, MRCP PhD, Principal Investigator — London School of Hygiene & Tropical Medicine, London, UK/Ifakara Health Research & Development Centre, Tanzania; Hassan Mshinda, PhD, Principal Investigator — Ifakara Health Research & Development Centre, Tanzania; Joanna RM Armstrong Schellenberg, PhD, Principal Investigator — London School of Hygiene & Tropical Medicine, London, UK/Ifakara Health Research & Development Centre, Tanzania; Pedro L Alonso, MD PhD, Principal Investigator — Hospital Clinic, Barcelona, Spain; Marcel Tanner, PhD, Principal Investigator — Swiss Tropical Institute, Basle, Switzerland
Locations (1):
- Ifakara Health Research & Development Centre, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Shamba D, Schellenberg J, Hildon ZJ, Mashasi I, Penfold S, Tanner M, Marchant T, Hill Z. Thermal care for newborn babies in rural southern Tanzania: a mixed-method study of barriers, facilitators and potential for behaviour change. BMC Pregnancy Childbirth. 2014 Aug 11;14:267. doi: 10.1186/1471-2393-14-267. PMID 25110173
- [Derived] Maokola W, Chemba M, Hamisi Y, Mrisho M, Shirima K, Manzi F, Masanja M, Willey B, Alonso P, Mshinda H, Tanner M, Schellenberg JR, Schellenberg D. Safety of sulfadoxine/pyrimethamine for intermittent preventive treatment of malaria in infants: evidence from large-scale operational research in southern Tanzania. Int Health. 2011 Sep;3(3):154-9. doi: 10.1016/j.inhe.2011.03.009. PMID 24038364
- [Derived] Shamba DD, Schellenberg J, Penfold SC, Mashasi I, Mrisho M, Manzi F, Marchant T, Tanner M, Mshinda H, Schellenberg D, Hill Z. Clean home-delivery in rural Southern Tanzania: barriers, influencers, and facilitators. J Health Popul Nutr. 2013 Mar;31(1):110-7. doi: 10.3329/jhpn.v31i1.14755. PMID 23617211
- [Derived] Schellenberg JR, Maokola W, Shirima K, Manzi F, Mrisho M, Mushi A, Alonso P, Mshinda H, Tanner M, Schellenberg DM. Cluster-randomized study of intermittent preventive treatment for malaria in infants (IPTi) in southern Tanzania: evaluation of impact on survival. Malar J. 2011 Dec 30;10:387. doi: 10.1186/1475-2875-10-387. PMID 22208409
- [Derived] Penfold S, Hill Z, Mrisho M, Manzi F, Tanner M, Mshinda H, Schellenberg D, Armstrong Schellenberg JR. A large cross-sectional community-based study of newborn care practices in southern Tanzania. PLoS One. 2010 Dec 21;5(12):e15593. doi: 10.1371/journal.pone.0015593. PMID 21203574
- See also: Intermittent Preventive Treatment in Infants (IPTi) Consortium — http://www.ipti-malaria.org/